CLINICAL TRIAL: NCT06551532
Title: An In-season Ecological Program Performed by Soccer Players Changes Pelvic Kinematics During Static, Linear Sprinting and Sport-specific Tasks: a Pilot Study on the Implication for Hamstring Injuries.
Brief Title: "Ecological Program Changes Pelvic Kinematics in Soccer Players: Pilot Study on Hamstring Injury Implications"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RX2 Sports and Health (Other)
Responsible Party: Principal Investigator, Andrea Astrella, Principal Investigator and PhD Candidate., RX2 Sports and Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RX2_EstudioHamstring_2024
Record Dates: First submitted 2024-08-07; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Anterior Pelvic Tilt; Sprint Kinematics
Keywords: Hamstring strain; Muscle Injury; Pelvic Tilt; Sprint Kinematics; Sprint Mechanics

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either an intervention group receiving the multicomponent intervention or a control group with no intervention, with both groups being monitored concurrently throughout the 6-week period.
Masking Description: In this study, both participants and researchers are aware of the group assignment. Participants know whether they are receiving the multicomponent intervention or are part of the control group. The researchers who administer the intervention and collect data are also aware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent Intervention Group (Experimental): Soccer players in the intervention group (IG) underwent a multimodal training program comprising 3 sessions per week for 6 weeks. All the soccer players in IG were allowed to continue their usual training (5 sessions per week) and matches (1 per week) at their clubs. The training program comprised both lumbopelvic training (foam rolling, manual therapy, mobility, posture, and strength training) and sprint technique components. The intervention included a total of 18 sessions of approximately 50 minutes each and sessions were supervised by 2 physiotherapists. During the 6 weeks of the intervention, participants performed the multicomponent program 3 times a week. Monday, Wednesday, and Friday were the chosen days for carrying out the training program, as Sunday was usually a game day.
  Interventions: Other: Multicomponent program
- Control Group (No Intervention): Soccer players in the control group (CG) were requested not to modify their established training routines during the entire 6-week period.

INTERVENTIONS:
Other: Multicomponent program — Lumbopelvic training (foam rolling, manual therapy, mobility, posture, and strength training) and sprint technique program.
  Arms: Multicomponent Intervention Group

SUMMARY:
The present pilot study aimed to investigate whether a 6-week multicomponent intervention, comprising a structural lumbopelvic and sprint technique program, could reduce anterior pelvic tilt in soccer players who regularly participated in soccer practice.

DETAILED DESCRIPTION:
This pilot study aimed to evaluate the impact of a 6-week multicomponent intervention combining lumbopelvic control exercises and running technique training on pelvis structure and lower limb kinematics in semi-professional soccer players. Seventeen players were randomly assigned to a control group (CG) or an intervention group (IG). Data on static anterior pelvic tilt (APT) and three-dimensional kinematics during high-speed running (HSR) and high-speed soccer running (HSSR) were collected before (PRE) and after (POST) the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for both groups were: (a) being between 18 and 40 years old, and (b) being available for their teams

Exclusion Criteria:

* Exclusion criteria for both groups included (a) not having suffered any musculoskeletal injuries in the previous 3 months and (b) not being involved in any additional strength program outside of their regular team training.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Anterior Pelvic Tilt (APT) Reduction. | Baseline (PRE) and immediately after 6 weeks of intervention (POST).
  The primary outcome measure is the reduction in static anterior pelvic tilt (APT) immediately after 6 weeks of the multicomponent intervention. APT is measured using a three-dimensional kinematic analysis during static and high-speed running tasks. The reduction in APT will be assessed before (PRE) and immediately after (POST) the intervention period to determine the effectiveness of the intervention in modifying pelvic alignment.

SECONDARY OUTCOMES:
biomechanical variables during high-speed running (HSR) and high-speed soccer running (HSSR) tasks | Baseline (PRE) and immediately after 6 weeks of intervention (POST).
  "This outcome measure assesses changes in specific biomechanical variables, including segment orientations (trunk, pelvis, femur, and tibia) relative to the sagittal plane, and joint angles (hip flexion and knee flexion) during high-speed running (HSR) and high-speed soccer running (HSSR) tasks. The study aims to evaluate the shift towards a more front-side oriented sprint technique model and the associated improvements in sprint performance time. Measurements will be taken using three-dimensional motion capture analysis to quantify the kinematic changes during HSR and HSSR."

CONTACTS AND LOCATIONS:
Locations (1):
- RX2 Sports and Health, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No